CLINICAL TRIAL: NCT01220479
Title: Impact of an Exercise Training Program on Bone Development and Cardiovascular Disease Risk Factors in Children With Type 1 Diabetes Mellitus
Brief Title: Exercise Training Intervention in Children With Type 1 Diabetes
Acronym: Diabex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Farpour-Lambert Nathalie, University Hospital of Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: snf n°63164
Record Dates: First submitted 2010-05-04; First posted 2010-10-14 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes, Bone mineral density, Growth; Cardiovascular diseases, Exercise, Training,; Child, Adolescent
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Healthy (No Intervention)
  Interventions: Behavioral: Exercise training program
- Control Diabetic (No Intervention)
  Interventions: Behavioral: Exercise training program
- Exercise Diabetic (Experimental)
  Interventions: Behavioral: Exercise training program
- Exercise Healthy (Experimental)
  Interventions: Behavioral: Exercise training program

INTERVENTIONS:
Behavioral: Exercise training program — Exercise Diabetic and Healthy groups perform a similar training program including two exercise sessions per week, of 90 minutes each, during 9 months (excluding holidays) under supervision by physical education teachers and pediatricians. Sessions comprise various weight-bearing activities: rope skipping, jumping, ball games and gymnastics.
  Control groups are relatively inactive.

SUMMARY:
Type 1 diabetes mellitus (T1DM) is associated with multiple co-morbidities, such as hypertension, dyslipidemia, coronary heart disease and osteoporosis. The foundation of these conditions lays in childhood. Exercise is known to have a positive influence on bone mineral density (BMD) and some impact on cardiovascular disease risk factors in healthy children, but little is known about these associations in children with T1DM.

The main purpose of this study is to assess the effects of a 9-month weight-bearing exercise training program on skeletal development in children with T1DM, compared to healthy subjects. The second aim is to evaluate whether the program influences also cardiovascular diseases risk factors.

This is a randomized controlled study incorporating 30 children with T1DM and 30 healthy children. Both groups are randomly divided (1:1) in an exercise or a control group: 1) exercise diabetic, 2) controls diabetic, 3) exercise healthy, 4) controls healthy.

Exercise groups participate to an identical weight-bearing exercise training program 2 x 90 minutes per week and controls are relatively inactive.

Main measures include: total body, lumbar spine and hip BMD by DXA, body fat and fat-free mass, bone biomarkers levels, resting and ambulatory blood pressure and fasting blood lipids.

ELIGIBILITY:
List of inclusion criteria for Type 1 diabetes patients:

1) disease for at least 1 year.

List of inclusion criteria for healthy subjects:

1) good general health and normal growth.

List of exclusion Criteria for all subjects:

1. presence of other chronic disease, including thyroid disease;
2. medications, hormones other than insulin, or calcium preparations taken in the preceding 6 months;
3. presence of nephropathy;
4. systemic disease or hospitalization for more than 2 weeks in the preceding year;
5. less than 6 menstrual cycles in the past year for post-menarche girls;
6. participation in competitive sport.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2001-09; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Bone mineral density and content | Baseline
  Assessment of bone mineral density (BMD) and content (BMC) at the whole body, hip and lumbar spine using DXA.
Bone mineral density and content | at 9 months
  Assessment of bone mineral density (BMD) and content (BMC) at the whole body, hip and lumbar spine using DXA.

SECONDARY OUTCOMES:
Anthropometrics | Baseline
  Body weight, height, body mass index and pubertal stage
Blood lipids levels | Baseline
  Fasting total cholesterol, LDL-Cholesterol, HDL-Cholesterol, triglycerides, lipoprotein (a), apolipoproteins A-I and B levels.
Physical activity | Baseline
  Physical activity level by questionnaire and accelerometer
Nutrition | Baseline
  Total energy, proteins, lipids, carbohydrates and calcium intakes using food records
Circulating bone biomarkers levels | Baseline
  Serum levels of beta-CrossLaps (CTX), N-MID-Osteocalcin (OC), N-Terminal Propeptide of Type I Collagen (PINP) and 25-OH-vitamin D (25-OH-D)
Glycated Haemoglobin | Baseline
  capillary HbA1c levels
Systemic blood pressure | Baseline
  Resting and 24-hour ambulatory systemic blood pressure monitoring
Body composition | Baseline
  Assessment of whole body and abdominal fat mass, and total fat-free mass using DXA.
Anthropometrics | at 9 months
  Body weight, height, body mass index and pubertal stage
Blood lipids levels | at 9 months
  Fasting total cholesterol, LDL-Cholesterol, HDL-Cholesterol, triglycerides, lipoprotein (a), apolipoproteins A-I and B levels.
Physical activity | at 9 months
  Physical activity level by questionnaire and accelerometer
Nutrition | at 9 months
  Total energy, proteins, lipids, carbohydrates and calcium intakes using food records
Circulating bone biomarkers levels | at 9 months
  Serum levels of beta-CrossLaps (CTX), N-MID-Osteocalcin (OC), N-Terminal Propeptide of Type I Collagen (PINP) and 25-OH-vitamin D (25-OH-D)
Glycated Haemoglobin | at 3 months
  capillary HbA1c levels
Glycated Haemoglobin | at 6 months
  capillary HbA1c levels
Glycated Haemoglobin | at 9 months
  capillary HbA1c levels
Systemic blood pressure | at 9 months
  Resting and 24-hour ambulatory systemic blood pressure monitoring
Body composition | at 9 months
  Assessment of whole body and abdominal fat mass, and total fat-free mass using DXA.

CONTACTS AND LOCATIONS:
Overall Officials: Farpour-Lambert Nathalie, PD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Maggio AB, Rizzoli RR, Marchand LM, Ferrari S, Beghetti M, Farpour-Lambert NJ. Physical activity increases bone mineral density in children with type 1 diabetes. Med Sci Sports Exerc. 2012 Jul;44(7):1206-11. doi: 10.1249/MSS.0b013e3182496a25. PMID 22246217